CLINICAL TRIAL: NCT05709366
Title: Knowledge, Beliefs and Attitudes of Greek Physiotherapist About the Using of Pain Neuroscience Education Program in Chronic Musculoskeletal Patients
Brief Title: Knowledge, Beliefs and Attitudes of Greek Physiotherapist About Pain Neuroscience Education
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantina Savvoulidou, Principal Investigator, University of Thessaly
Other Study IDs: N7
Record Dates: First submitted 2023-01-20; First posted 2023-02-02 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Pain Neuroscience Education; Chronic Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An e-survey study will be carried out based on Checklist for Reporting Results of 52 Internet E-Surveys (CHERRIES)". The purpose of this study is to investigate the knowledge, beliefs and behaviour of Greek physiotherapists regarding the pain neuroscience education program (PNE) as an intervention in patients with chronic musculoskeletal pain.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

What physiotherapists know about a PNE program; What physiotherapists believe about the using of a PNE program in patients with chronic musculoskeletal pain? Whether and how often they use a PNE program in patients with chronic musculoskeletal pain? What are the barriers of using PNE in patients with chronic musculoskeletal pain?

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapists who are member of Panhellenic Association of Physiotherapist in Greece, with active clinical practice in Greece and clinical experience in musculoskeletal disorders (>12 months).

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physiotherapists with chronic musculoskeletal experience and clinical practice in Greece
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Demographic characteristics | Baseline
  Questions will include participants' demographic characteristics (e.g. gender, age), 2) the setting where they practice their profession (e.g. hospital, private physiotherapy clinic), 3) level of education (e.g. BSc, MSc), 5) their years of practice, 6) seminars or training programs they have attended regarding pain neuroscience education.
Knowledge related to Pain Neuroscience Education | Baseline
  A question about how much do they know about Pain Neuroscience Education using a 10-point Likert scale, where 0=I don't know anything about the concept and 10=I have comprehensive knowledge on the concept."
Beliefs related to Pain Neuroscience Education | Baseline
  A question about how much do they believe a Pain Neuroscience Education is useful as an intervention in chronic musculoskeletal patients, using a 6-point Likert scale, where 0=completely disagree and 10=completely agree.
Attitudes related to Pain Neuroscience Education | Baseline
  A question about the application of a Pain Neuroscience Education as an intervention in chronic musculoskeletal patients, using a 6-point Likert scale, where 0=completely disagree and 10=completely agree.
Barriers related to Pain Neuroscience Education | Baseline
  5 statements with specific barriers for Pain Neuroscience Education using a 6-point Likert scale, where 0=completely disagree and 10=completely agree and an open question about other barriers.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Kapreli, PhD, Study Director — University of Thessaly
Locations (1):
- University of Thessaly, Lamia, Greece